CLINICAL TRIAL: NCT02307526
Title: Acetylcholinesterase Inhibition: A Novel Approach in the Treatment of Orthostatic Hypotension in Spinal Cord Injury
Brief Title: Acetylcholinesterase Inhibition and Orthostatic Hypotension in SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Specialist, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEC-11-04
Record Dates: First submitted 2014-05-21; First posted 2014-12-04 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hypotension, Postural
Keywords: Hypotension, Postural
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Pyridostigmine Bromide; Tilt-Table Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Cord Injury (Experimental): After being transferred onto a tilt table, subject with complete SCI will lie in a rested, supine position in which the study drug, pyridostigmine bromide (60 mg) will be administered at the 30 minute time point. Following the administration of the study drug, the subject will remain in the supine position for an additional 30 minutes until the tilting protocol commences.
  Interventions: Drug: Pyridostigmine Bromide; Device: Tilt table test

INTERVENTIONS:
Drug: Pyridostigmine Bromide — After being transferred onto a tilt table, subject will lie in a rested, supine position in which the study drug, pyridostigmine bromide will be administered at the 30 minute time point. Following the administration of the study drug, the subject will remain in the supine position for an additional 30 minutes until the tilting protocol commences.
  Other Names: Brand Name: Mestinon
Device: Tilt table test — After 60 minutes in supine resting position, a progressive head-up tilt will be utilized in which the table will be adjusted to 15°, 25°, 35° for 5 minutes at each angle and then maintained at 45° for 45 minutes or until the subjects experiences symptoms of compromised cerebral blood flow, which include, but are not limited to, light headedness, blurry vision, dizziness and nausea.
  Other Names: Upright tilt testing

SUMMARY:
Due to de-centralized cardiovascular control, persons with spinal cord injury (SCI) experience blood pressure (BP) dysregulation which manifests in chronic hypotension with exacerbation during orthostatic positioning. Although many individuals with SCI remain asymptomatic to hypotension and orthostatic hypotension (OH), we recently reported reduced memory and marginally reduced attention and processing speed in hypotensive individuals with SCI compared to a normotensive cohort. Thus, we believe that treatment of overtly asymptomatic hypotension and OH in the SCI population is clinically warranted. Currently the FDA has approved only midodrine hydrochloride for the treatment of dizziness associated with OH and proof of efficacy is limited. Acetylcholinesterase inhibition for treatment of OH is a novel concept and has gained recent recognition in models of neurogenic OH (multiple system atrophy; pure autonomic failure, diabetic neuropathy). The physiological rationale of this concept is unique: acetylcholine (AcH) is the pre-ganglionic neurotransmitter of the sympathetic nervous system. Inhibition of acetylcholinesterase will limit the breakdown of AcH thereby facilitating vascular adrenergic tone and peripheral vasoconstriction. Acetylcholinesterase inhibition has been reported to be efficacious in models of both pre-ganglionic (multiple system atrophy) and post-ganglionic (pure autonomic failure, diabetic neuropathy) origin and persons with SCI reflect a model of a preganglionic disorder. In theory, if an individual has a complete autonomic lesion, acetylcholinesterase inhibition would not be expected to improve orthostatic BP because little/no neural traffic would be transmitted to the pre-synapse. However, individuals with an incomplete autonomic lesion may benefit from this class of agent. Researchers are currently investigating the orthostatic BP effects of acetylcholinesterase inhibition with pyridostigmine bromide (60 mg) in 10 individuals with SCI.

DETAILED DESCRIPTION:
Due to de-centralized cardiovascular control, persons with spinal cord injury (SCI) experience blood pressure (BP) dysregulation which manifests in chronic hypotension with exacerbation during orthostatic positioning. Although many individuals with SCI remain asymptomatic to hypotension and orthostatic hypotension (OH), we recently reported reduced memory and marginally reduced attention and processing speed in hypotensive individuals with SCI compared to a normotensive cohort. Thus, we believe that treatment of overtly asymptomatic hypotension and OH in the SCI population is clinically warranted. Currently the FDA has approved only midodrine hydrochloride for the treatment of dizziness associated with OH and proof of efficacy is limited. Acetylcholinesterase inhibition for treatment of OH is a novel concept and has gained recent recognition in models of neurogenic OH (multiple system atrophy; pure autonomic failure, diabetic neuropathy). The physiological rationale of this concept is unique: acetylcholine (AcH) is the pre-ganglionic neurotransmitter of the sympathetic nervous system. Inhibition of acetylcholinesterase will limit the breakdown of AcH thereby facilitating vascular adrenergic tone and peripheral vasoconstriction. Acetylcholinesterase inhibition has been reported to be efficacious in models of both pre-ganglionic (multiple system atrophy) and post-ganglionic (pure autonomic failure, diabetic neuropathy) origin and persons with SCI reflect a model of a preganglionic disorder. In theory, if an individual has a complete autonomic lesion, acetylcholinesterase inhibition would not be expected to improve orthostatic BP because little/no neural traffic would be transmitted to the pre-synapse. However, individuals with an incomplete autonomic lesion may benefit from this class of agent. Researchers are currently investigating the orthostatic BP effects of acetylcholinesterase inhibition with pyridostigmine bromide (60 mg) in 10 individuals with SCI. The primary objectives of this study are to compare the BP response to head-up tile (HUT: 45°) between no-drug and drug (pyridostigmine 60 mg) in individuals with SCI with documented OH; and to compare the orthostatic BP responses following drug in individuals with SCI.

Subjects will be tested on two separate days. On day 1 of testing, subjects will be transferred onto a tilt table and will remain in the supine position for the entirety of the test. During the first 60 minutes the subject will remain at the resting supine position.

Following the 60 minute resting position, a progressive head-up tilt will be utilized in which the table will be adjusted to 15°, 25°, 35° for 5 minutes at each angle and then maintained at 45° for 45 minutes or until the subjects experiences symptoms of compromised cerebral blood flow, which include, but are not limited to, light headedness, blurry vision, dizziness and nausea.

On day 2 of testing, the protocol will be duplicated with the exception of drug administration. 60 mg of the study drug, pyridostigmine will be administered at the 30 minute mark of the resting supine position. Data for heart rate and blood pressure will be monitored continuously during the progressive HUT maneuver and will be recorded at 10 minute intervals during the 45° HUT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Spinal cord injury with American Spinal Injury Association Impairment Scale (AIS) level of Grade A, B, C or D 9non-ambulatory)
* Neurological level of injury C3-T2
* Duration of injury greater than 1 year

Exclusion Criteria:

* Currently taking medications with known blood pressure raising or lowering effects.
* Taking over-the-counter medications for allergies or cold symptoms 24-hours prior to testing.
* I have a C3 level of injury and I am ventilator dependent.
* History of cardiovascular arrhythmias (especially slow heart rate, less than 45 bpm), block in the electrical signal within the heart, cardiac arrest.
* History of convulsions or seizures.
* Currently taking medication to treat active asthma.
* Thyroid problems.
* Current smoker.
* Known coronary heart and/or artery disease.
* High blood pressure
* Diabetes
* Current illness or infection
* Major surgery in the last 30 days
* Hypersensitivity to pyridostigmine, bromides, or any component of the formulation; (as determined by review of known drug allergies reported in the medical history intake form and confirmed by the study physician)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M. Wecht, EdD, Principal Investigator — James J. Peters VAMC
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Injury: 10 individuals with spinal cord injury (SCI: C4-C7) were recruited.
Period: Day 1 - No Drug
Arm/Group | Spinal Cord Injury
Started | 10
Completed | 10
Not Completed | 0
Period: Day 2 - 60 mg of Pyridostigmine
Arm/Group | Spinal Cord Injury
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Spinal Cord Injury: Ten individuals with SCI (C4-C7) were recruited.
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Time Frame: Average systolic blood pressure of 10 minutes supine rest before pyridostigmine and after 45 minutes at 45 degrees after pyridostigmine administration compared to 10 minutes supine rest before tilt and at 45 degrees during no-drug head-up tilt maneuver.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- NO Drug: Following the 60 minute resting position, a progressive head-up tilt will be utilized in which the table will be adjusted to 15°, 25°, 35° for 5 minutes at each angle and then maintained at 45° for 45 minutes or until the subjects experiences symptoms of compromised cerebral blood flow, which include, but are not limited to, light headedness, blurry vision, dizziness and nausea.
Arm/Group | Pyridostigmine Bromide | NO Drug
Number analyzed (Participants) | 10 | 10
mm Hg
  Supine Systolic Blood Pressure | 97 (11) | 103 (14)
  45 degree Head-up Tilt Systolic Blood Pressure | 90 (18) | 88 (12)

2. Primary Outcome: Diastolic Blood Pressure
Time Frame: Average diastolic blood pressure of 10 minutes supine rest before pyridostigmine and after 45 minutes at 45 degrees after pyridostigmine administration compared to 10 minutes supine rest before tilt and at 45 degrees during no-drug head-up tilt maneuver.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pyridostigmine Bromide | NO Drug
Number analyzed (Participants) | 10 | 10
mm Hg
  Supine Diastolic Blood Pressure | 64 (6) | 66 (10)
  45 degree Head-up Tilt Diastolic Blood Pressure | 64 (11) | 63 (7)

3. Primary Outcome: Heart Rate
Time Frame: Average heart rate of 10 minutes supine rest before pyridostigmine and after 45 minutes at 45 degrees following pyridostigmine administration compared to 10 minutes supine rest before tilt and at 45 degrees during no-drug head-up tilt maneuver.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Pyridostigmine Bromide | NO Drug
Number analyzed (Participants) | 10 | 10
bpm
  Supine Heart Rate | 52 (6) | 55 (10)
  45 degree Head-up Tilt Heart Rate | 66 (12) | 72 (13)

ADVERSE EVENTS:
Time Frame: 80 minuets after pyridostigmine administration to 200 minuets after pyridostigmine administration.
Groups:
- Day 1 - No Drug: Following the 60 minute resting position, a progressive head-up tilt will be utilized in which the table will be adjusted to 15°, 25°, 35° for 5 minutes at each angle and then maintained at 45° for 45 minutes or until the subjects experiences symptoms of compromised cerebral blood flow, which include, but are not limited to, light headedness, blurry vision, dizziness and nausea.
- Day 2 - Pyridostigmine Bromide: After being transferred onto a tilt table, subject will lie in a rested, supine position in which the study drug, pyridostigmine bromide 60 mg will be administered at the 30 minute time point. Following the administration of the study drug, the subject will remain in the supine position for an additional 30 minutes until the tilting protocol commences.
Arm/Group | Day 1 - No Drug | Day 2 - Pyridostigmine Bromide
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 1 - No Drug (N=10) | Day 2 - Pyridostigmine Bromide (N=10)
Drug Side Effect (Nervous system disorders) | 0 (0) | 1 (1) — One participant reported increased sweating and salivation following pyridostigmine administration.
Overheating (Nervous system disorders) | 0 (0) | 1 (1) — One subject terminated head-up tilt intervention due to overheating.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No